CLINICAL TRIAL: NCT06327412
Title: Effects of Hospital-Based Aerobic Exercise Therapy on Exercise Capacity, Body Composition, Functional Level and Quality of Life in Patients With Primary Lower Extremity Lymphedema; Prospective Randomized Controlled Single Blind Trial
Brief Title: The Effects of Aerobic Exercise in Patients With Primary Lower Extremity Lymphedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, professor doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KayseriCHLYMP01
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Primary Lymphedema; Aerobic Exercise
Keywords: primary lymphedema; aerobic execise; Cardiopulmonary Exercise Test; cardiopulmonary rehabilitation
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: A total of 35 patients with primary stage 2 and 3 lower extremity lymphedema, aged 18-65, who apply to the lymphedema outpatient clinic and meet the criteria of the International Society of Lymphology, will be included. Patients participating in the study will be randomized into 2 groups: aerobic exercise group (Group 1) and home exercise group (Group 2). According to randomization, 18 patients will be included in one group and 17 patients in the other.
  Cardiopulmonary exercise test (CPET), 30-second-stand-sit test (30s-CST), 6-minute walk test (6MWT), Lymphedema Circumference and Volume Measurement, Bioimpedance Measurement, Lower Extremity Functional Scale (LEFS), Lymphedema Life Impact Scale ( LLIC), Hospital Depression and Anxiety Scale (HADS), Numerical Rating Scale (NRS) forms will be filled in the cardiopulmonary rehabilitation unit of Kayseri City Hospital in the 0th, 4th and 16th weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital Exercise Group (Active Comparator): According to the Cardiopulmonary Exercise test (CPET), the patients should exercise on the treadmill (5 minutes warm-up, 30 minutes exercise, 5 minutes cool-down) for 40 minutes (5 minutes warm-up, 30 minutes exercise, 5 minutes cool-down) at an exercise intensity of 50-60% of the individually recorded VO2 max (the maximum amount of oxygen that an individual can utilize during intense or maximal exercise) level in the patients. Aerobic exercise therapy will be organized to include treadmill.
  Interventions: Other: Aerobic exercise on the treadmill
- Home Exercise Group (Placebo Comparator): Patients will be asked to walk 40 minutes a day, 5 days a week, for 4 weeks. Training will be given for the first session in the hospital to ensure that the patient's walking pace is between 12-13 RPE (The Borg Rating of Perceived Exertion) according to the Modified Borg scale.
  Interventions: Other: Walking between 12-13 RPE (The Borg Rating of Perceived Exertion) according to the Modified Borg Scale

INTERVENTIONS:
Other: Aerobic exercise on the treadmill — According to the cardiopulmonary exercise (CPET) test, 40 minutes (5 minutes warm-up, 30 minutes exercise, 5 minutes cool-down) at an exercise intensity of 50-60% of the VO2 max (the maximum amount of oxygen that an individual can utilize during intense or maximal exercise) level recorded individually in patients, 5 days a week for 4 weeks.Both patient groups will be given lymphedema-specific remedial exercise program training. Anatolian Lymphedema Association lower extremity lymphedema exercise sheets will be delivered to the patients in writing, and training on exercise practices will be given face to face as a session by a physiotherapist at the physical therapy lymphedema outpatient clinic. Patients will be asked to perform these exercises daily as stated in the leaflet and in the number of repetitions. Patients will be given an exercise diary to ensure their compliance with exercise and will be asked to mark this form daily
  Arms: Hospital Exercise Group
Other: Walking between 12-13 RPE (The Borg Rating of Perceived Exertion) according to the Modified Borg Scale — He/she will be asked to walk 40 minutes a day, 5 days a week, for 4 weeks. Training will be given for the first session in the hospital to ensure that the patient's walking pace is between 12-13 RPE according to the Modified Borg scale.Both patient groups will be given lymphedema-specific remedial exercise program training. Anatolian Lymphedema Association lower extremity lymphedema exercise sheets will be delivered to the patients in writing, and training on exercise practices will be given face to face as a session by a physiotherapist at the physical therapy lymphedema outpatient clinic. Patients will be asked to perform these exercises daily as stated in the leaflet and in the number of repetitions. Patients will be given an exercise diary to ensure their compliance with exercise and will be asked to mark this form daily.Treatment compliance will be increased by making weekly phone calls to patients in order to increase treatment compliance and evaluate compliance.
  Arms: Home Exercise Group

SUMMARY:
Our aim in this study is to evaluate the effects of lymphedema on exercise capacity, body composition, functional level and quality of life in lymphedema patients with primary lower extremity involvement.

DETAILED DESCRIPTION:
Male and female patients aged 18-65, who applied to Kayseri City Hospital's Department of Physical Medicine and Rehabilitation (PMR), lymphedema outpatient clinic between September 2023 and September 2024 due to lower extremity edema, will be included in this study. Lymphedema was diagnosed by clinical and/or imaging methods (lower extremity circumference difference measurements, venous Doppler ultrasonography, lymphoscintigraphy), evaluated by an PMR specialist physician, phase 1 decongestive treatment was applied within the last month, stage 2-3 lower legs using Class 3 compression stockings were used. Patients with extremity lymphedema will be included. Our study is a prospective, randomized controlled, single-blind clinical trial. In our study, survey forms will be filled out by a researcher who is blind to the applied tests and study groups. Patients will be divided into 2 groups according to computerized randomization.

Demographic data such as age, gender, occupational status, education level, marital status of the patients whose verbal and written consent was obtained; Height, body weight, body mass index, smoking-alcohol use, medications used and additional diseases will be questioned and recorded in their files.

The lower extremity circumference of the patients will be measured with a flexible standard tape measure that is 150 cm long, 1 cm wide and spaced one cm apart. Measurements will be marked including the metatarsophalangeal joint, the middle of the dorsum of the foot, the ankle, and the end of the thigh at 4 cm intervals from this area. Circumference measurement from the marked points will be repeated twice each time by a physiatrist blinded to the study, and the average of the two measurements will be taken. These measurements will be repeated at the beginning of the study and at weeks 4 and 16.

The total extremity volume will be determined by calculating the data obtained from the circumference measurement with the Frustum formula, which is used to indirectly determine the extremity volume. The difference between both lower extremities before and after treatment will be determined. These evaluations will be repeated at the beginning of the study and at weeks 4 and 16.

The body extracellular fluid ratio will be determined by the bioelectrical impedance method using a body composition analyzer in which the impedance in the tissues is analyzed by applying a low level of electric current to the body. This measurement will be repeated at the beginning of the study and at weeks 4 and 16.

CPET test will be performed in patients to evaluate their aerobic exercise capacity. CPET tests will be applied with a device in the Cardiopulmonary Rehabilitation Unit of Kayseri City Hospital Physical Therapy and Rehabilitation Department. All patients will be informed about the exercise test before the test. Patients will undergo a detailed physical examination, height, body weight, body mass index, heart rate, blood pressure will be measured and evaluated by taking a baseline ECG. The change in the patient's exercise capacity will be evaluated at the 0th, 4th and 16th weeks according to the VO2 max (the maximum amount of oxygen that an individual can utilize during intense or maximal exercise) value in the CPET test. The CPET test and questionnaires administered to all patients who complete the treatment before treatment will be re-evaluated at the 4th and 16th weeks.

In Group 1 (Hospital-based aerobic exercise group), patients were given 40 minutes (5 minutes warm-up, 30 minutes exercise, 5 minutes exercise) for 4 weeks, 5 days a week, at an exercise intensity of 50-60% of the VO2 max level recorded individually in the patients according to the CPET test. Aerobic exercise therapy will be organized to be applied on a treadmill (in the form of a cooling down).

In Group 2 (Home-based exercise group), patients will be asked to walk 40 minutes a day, 5 days a week, for 4 weeks. Training will be given for the first session in the hospital to ensure that the patient's walking pace is between 12-13 RPE (The Borg Rating of Perceived Exertion) according to the Modified Borg scale.

Both patient groups will be given lymphedema-specific remedial exercise program training. Anatolian Lymphedema Association lower extremity lymphedema exercise sheets will be delivered to the patients in writing, and training on exercise practices will be given face to face as a session by a physiotherapist at the physical therapy lymphedema outpatient clinic. Patients will be asked to perform these exercises daily as stated in the leaflet and in the number of repetitions. Patients will be given an exercise diary to ensure their compliance with exercise and will be asked to mark this form daily. In the home exercise group, treatment compliance will be increased by making weekly phone calls to patients in order to increase treatment compliance and evaluate compliance.

Before the treatment, at the end of the 4-week treatment and at the 16th week, the patients had 30-second sit-to-stand test (30s-CST), 6-minute walk test (6MWT), Circumference-volume and bioimpedance measurement, Lower Extremity Functional Scale (LEFS), Lymphedema Life Impact. Scale (LLIC), Hospital Depression and Anxiety scale (HADS), Numerical Rating Scale (NRS) forms will be filled out.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed complete decongestive therapy (CBT) Phase 1 treatment within the last 1 month, use Class 3 compression garments, and are scheduled for CBT Phase 2 treatment.
* Patients with stage 2-3 unilateral or bilateral primary lymphedema with lower extremity involvement
* Women and men aged 18-65
* Patients who agreed to participate in the study and received written voluntary consent form.

Exclusion Criteria:

* Patients who do not agree to participate in the study
* Patients without cooperation and compliance
* Presence of phlebo edema, lipedema, cellulitis, lymphocele
* History of lower extremity venous system disease
* Presence of acute infection
* History of malignancy
* Presence of acute/chronic lung disease (history of acute pulmonary embolism, acute bronchial asthma attack, chronic interstitial lung disease)
* Chronic liver failure
* Renal dysfunction
* Uncontrolled hypertension and diabetes mellitus
* Presence of orthopedic disease that may prevent walking (joint limitation, ankylosis, amputation)
* Use of medications known to affect physical performance, heart rate or metabolism (including Beta blockers)
* Patients who have been included in the CPR (Cardiopulmonary resuscitation) program in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
30-second sit-stand test (30-s chair-stand test, 30s-CST) | week 0, 4th week, 16th week
  It is a test with proven validity and reliability that evaluates the patient's sit-to-stand activity, lower extremity strength and dynamic balance. The patient's sitting height is approximately 43 cm on a chair without arms; The patient is asked to sit with his back straight and straight, his arms crossed in front, his feet on the floor, and then he is asked to sit and stand within 30 seconds. The number of times he sits and stands gives the score of the test.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | week 0, 4th week, 16th week
  It is a non-invasive procedure that evaluates the individual's capacity during dynamic exercise and provides diagnostic and prognostic information. CPET is based on the investigation of the respiratory system, cardiovascular system and cellular response to exercise performed under controlled metabolic conditions. It allows detailed, holistic physiological evaluation of the organs involved in exercise. Patients should be informed that they should wear comfortable clothes, stop eating and drinking 3 hours before the exercise test, and avoid smoking and drinking alcohol. Before the test, patients should be informed about the test, a detailed physical examination should be performed, and contraindications, if any, should be determined
6-minute walk test (6MWT) | week 0, 4th week, 16th week
  It is a frequently used test in cardiopulmonary rehabilitation to monitor exercise capacity and treatment effectiveness. The patient should rest by sitting in a chair for 15 minutes before the test and wear appropriate shoes and comfortable clothing. Calculate the distance walked by the patient at their own walking pace in 6 minutes, preferably in a 30-meter long corridor. If the patient's O2 saturation (sO2) is <88%, the test should be performed with O2 support.
Circumference and volume measurement | week 0, 4th week, 16th week
  Circumference measurement, which is made by taking measurements from certain points of the extremity, is one of the frequently used, easy-to-apply methods to determine the extremity volume and used to determine the severity of lymphedema. When measuring the circumference, the position of the extremity should be constant, and the same position should be maintained for the opposite side or repeated measurements, and the intervals used should be equal. The data obtained from the circumference measurement is Frustum formula (Frustum Formula V= [ h x (R12+R1.R2+R22)] / (12 x π) VT (Leg volume) = V1+........Vn [V: volume, h: Range used in circumference measurement, R1: Base circumference measurement of the conical segment, R2: upper circumference measurement of the conical segment, VT: Leg volume, n: Number of conical segments.
Bioimpedance measurement | week 0, 4th week, 16th week
  Bioimpedance is defined as the body's resistance to applied electrical current. Estimates the extracellular fluid volume by measuring the bioimpedance created in the tissue by the alternating current transmitted to the extremity.
Lower Extremity Functional Scale (LEFS) | week 0, 4th week, 16th week
  Developed to evaluate individuals' lower extremity functions, abilities and activity limitations, and validated in Turkish; The scale consists of 20 items and there are 5 options for each question (0: extreme difficulty or inability to perform the activity, 1: quite a difficulty, 2: moderate difficulty, 3: some difficulty, 4: no difficulty). In the total score ranging from 0 to 80, higher scores indicate better functional status.
Lymphedema Life Impact Scale (LLIC) | week 0, 4th week, 16th week
  Developed specifically for lymphedema, it is a comprehensive scale used for lymphedema in both the upper and lower extremities. It consists of 18 items, 8 of which evaluate physical, 4 psychosocial, and 6 functional problems. High scores on the scale, which has a score between 1 and 5 for each item, indicate that the limitation in the relevant function is high. The scale, which questions the incidence of infection, which is a common and important complication in lymphedema, differs from other scales used in lymphedema in this respect.
Hospital Anxiety and Depression Scale (HADS) | week 0, 4th week, 16th week
  It is very important to recognize psychiatric disorders in people with physical illnesses. Psychiatric disease is not diagnosed with this test. It is a screening test that non-psychiatric physicians can also use in their work and clinical settings. HADS was designed to screen for anxiety and depression in people with physical illnesses. The cutoff score for HADS, depression and anxiety subscales is ≥ 8. The validity of the HAD Turkish translation was made by Aydemir et al. The survey includes seven questions for anxiety and seven questions for depression and takes 2-5 minutes to complete. 8-10; light, 11-14; middle, 15-21; is classified as severe.
Numerical Rating Scale (NRS) | week 0, 4th week, 16th week
  Used as a measure of pain intensity in adults. 0; no pain, 10; It is the strongest pain felt

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gül Ülkü Demir, MD, Study Director — Kayseri City Hospital; Firdevs Akdeniz Çınar, Principal Investigator — Health Sciences University, Kayseri Medical Faculty
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adachi H. Cardiopulmonary Exercise Test. Int Heart J. 2017 Oct 21;58(5):654-665. doi: 10.1536/ihj.17-264. Epub 2017 Sep 30. PMID 28966333
- [Background] Hamilton DM, Haennel RG. Validity and reliability of the 6-minute walk test in a cardiac rehabilitation population. J Cardiopulm Rehabil. 2000 May-Jun;20(3):156-64. doi: 10.1097/00008483-200005000-00003. PMID 10860197
- [Background] Sakamoto M, Suematsu Y, Yano Y, Kaino K, Teshima R, Matsuda T, Fujita M, Tazawa R, Fujimi K, Miura SI. Depression and Anxiety Are Associated with Physical Performance in Patients Undergoing Cardiac Rehabilitation: A Retrospective Observational Study. J Cardiovasc Dev Dis. 2022 Jan 11;9(1):21. doi: 10.3390/jcdd9010021. PMID 35050231
- [Background] Verbrugghe J, Agten A, Stevens S, Hansen D, Demoulin C, O Eijnde B, Vandenabeele F, Timmermans A. Exercise Intensity Matters in Chronic Nonspecific Low Back Pain Rehabilitation. Med Sci Sports Exerc. 2019 Dec;51(12):2434-2442. doi: 10.1249/MSS.0000000000002078. PMID 31269004